CLINICAL TRIAL: NCT06433817
Title: The Clinical Research of Spectral CT in Radiotherapy for Cervical Cancer
Brief Title: Spectral CT in Radiotherapy for Cervical Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SPRTCC-Trial
Record Dates: First submitted 2024-05-08; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer; Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Spectral computed tomography scan — Spectral CT scans acquisition performed during the arterial phase and venous phase for cervical cancer

SUMMARY:
The purpose of this study was to explore the potential application of spectral CT for radiotherapy in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were confirmed cervical cancer by pathology
2. patients were treated with concurrent chemoradiotherapy
3. Spectral CT scans acquisition performed during the arterial phase and venous phase
4. All the patients underwent a 18F-FDG PET/CT before treatment

Exclusion Criteria:

1. CT without spectral scans
2. History of allergy to intravenous contrast
3. Pregnant or potentially pregnant female subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with newly stablished diagnosis of cervical cancer complying with selection criteria for cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-22 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of spectral CT derived data with response evaluation in cervical cancer | through study completion, an average of 2 year
  To evaluate the tumor response of using quantitative parameters in spectral CT for cervical cancer patients according to RECIST 1.1

SECONDARY OUTCOMES:
Identifying metastatic lymph nodes in cervical cancer with spectral CT | through study completion, an average of 2 year
  To evaluate the diagnostic performances of using spectral CT for identifying metastatic lymph nodes in patients with cervical cancer
Application of energy spectrum CT in brachytherapy of cervical cancer | through study completion, an average of 2 year
  The ability to reduce metal artifact and assist in target delineation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No